CLINICAL TRIAL: NCT07020923
Title: A Study Evaluating Monthly (Every 4 Weeks) Dosing of Atacicept in Patients With IgAN
Brief Title: Monthly Dosing of Atacicept in IgAN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VT-001-0020
Record Dates: First submitted 2025-05-13; First posted 2025-06-13 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: IgA Nephropathy (IgAN); Berger Disease
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — TACI receptor-IgG Fc fragment fusion protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Atacicept Arm 1 (Experimental): Atacicept dose A administered subcutaneous (sc) injection monthly
  Interventions: Drug: Atacicept
- Atacicept Arm 2 (Experimental): Atacicept dose B administered subcutaneous (sc) injection monthly
- Atacicept Arm 3 (Experimental): Atacicept dose C administered subcutaneous (sc) injection monthly
- Atacicept Arm 4 (Experimental): Atacicept dose D administered subcutaneous (sc) injection weekly
- Atacicept Arm 5 (Experimental): Atacicept dose E administered subcutaneous (sc) injection weekly for 24 weeks, followed by monthly sc injections

INTERVENTIONS:
Drug: Atacicept — Drug: Atacicept
  Other Names: VT-001
  Arms: Atacicept Arm 1

SUMMARY:
This is a Phase 2, open-label, multicenter, randomized study comprising parallel groups of participants receiving weekly and/or monthly doses of atacicept

DETAILED DESCRIPTION:
This Phase 2 study is to explore the effectiveness, safety and tolerability of different dosing regimens of atacicept. Regimens include monthly and weekly dosing.

ELIGIBILITY:
Inclusion Criteria:

* Must have the ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study assessments
* Adult male or female of ≥18 years of age, or as per country specific legally or nationally recognized adult age, who provides written informed consent prior to performing any study assessments
* Diagnosis of IgAN as demonstrated by renal biopsy conducted within 10 years
* Total urine protein excretion ≥0.75 g per 24-hour or urine protein-to-creatinine ratio (UPCR) ≥0.75 mg/mg based on a 24-hour urine sample
* eGFR ≥30 mL/min/1.73 m2 at screening, as per the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI)
* On a stable prescribed regimen of RASi (angiotensin converting enzyme inhibitor or angiotensin II receptor blocker) for at least 8 weeks that is at the maximum labeled or tolerated dose at screening and from screening to study Day 1

Exclusion Criteria:

* IgAN secondary to another condition (eg, liver cirrhosis), or other causes of mesangial IgA deposition including IgA vasculitis (ie, Henoch-Schonlein purpura), systemic lupus erythematosus, dermatitis herpetiformis, ankylosing spondylitis
* Evidence of rapidly progressive glomerulonephritis (loss of ≥50% of eGFR within 3 months of screening)
* Evidence of nephrotic syndrome within 6 months of screening (serum albumin <3.0 g/dL in association with UPCR >3.5 mg/mg)
* Renal or other organ transplantation prior to or expected during the study, with the exception of corneal transplants
* Concomitant chronic renal disease in addition to IgAN (eg, diabetic nephropathy, primary focal segmental glomerulosclerosis, membranous nephropathy, C3 glomerulopathy, lupus nephritis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of atacicept on Gd-IgA1 in patients with IgAN | Up to 24 weeks
  Gd-IgA1 levels through Week 24

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of atacicept at different dosing regimensT | Baseline until end of study up to Week 24
  Incidence of treatment emergent reported Adverse Events (AE)
To evaluate the effect of atacicept on serum immunoglobulins (IgA) | 24 Weeks
  IgA levels through Week 24
To evaluate the effect of atacicept on serum immunoglobulins (IgG) | 24 Weeks
  IgG levels through Week 24
To evaluate the effect of atacicept on serum immunoglobulins (IgM) | 24 Weeks
  IgM levels through Week 24
To evaluate serum PK of atacicept | Baseline until end of study up to Week 24
  Serum concentration of atacicept

CONTACTS AND LOCATIONS:
Overall Officials: Zeeshan Khawaja, Study Director — Vice President, Clinical Development
Locations (1):
- Vera Therapeutics, Brisbane, California, United States

REFERENCES:
- See also: Vera Therapeutics, Inc Company Website — http://www.veratx.com